CLINICAL TRIAL: NCT01107132
Title: Blood-retinal Barrier Imaging in Type 2 Diabetes Mellitus: a Window for Blood-brain Barrier Breakdown and Neuropsychiatric Sequela
Brief Title: Blood-retinal Barrier Imaging and Neuropsychiatric Sequela in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Hadar Shalev, M.D, Soroka University Medical Center
Other Study IDs: SOR495710ctil
Record Dates: First submitted 2010-04-18; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Type 2 Diabetes Mellitus; Non-Proliferative Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — • Fluorescein Angiography
  1. Investigation and documentation of the retinal and choroidal vascular systems integrity by intravenous administration of sodium fluorescein
  2. FA images are recorded in a central database with restricted accesses and are routinely analyzed by the eye specialist
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetic Retinopathy: T2DM Patient suffering from Non-Proliferative Diabetic Retinopathy (NPDR), Proliferative Diabetic Retinopathy (PDR) and Diabetic Macular Edema (DME)

SUMMARY:
In Type 2 Diabetes mellitus patients we will:

1. quantify vasculopathy and blood-retinal barrier (BRB) leakage
2. measure blood-brain barrier (BBB) permeability and neuroanatomical changes
3. correlate BRB pathology with BBB breakdown, inflammatory markers and neuropsychiatric sequela

ELIGIBILITY:
Inclusion criteria:

1. T2DM Patient suffering from Non-Proliferative Diabetic Retinopathy (NPDR), Proliferative Diabetic Retinopathy (PDR) and Diabetic Macular Edema (DME) who are in the clinical database of the ophthalmologic department , above 18 years old at the time of diagnosis and underwent FA examination in the past three years
2. Patients which their medical records are available via a computerized data base

Control group:

1. T2DM patients who are in the clinical database of the ophthalmologic department
2. Above 18 years old at the time of diagnosis
3. Underwent FA examination in the past three years and their examination was interpreted as "normal", i.e. without suspected diabetic retinopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes Mellitus Patient suffering from Non-Proliferative Diabetic Retinopathy (NPDR), Proliferative Diabetic Retinopathy (PDR) and Diabetic Macular Edema
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Shalev, M.D, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel